209713

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for A Randomized, Open-Label, Single Dose, Four-Period Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants |
| <b>Compound Number</b> | : | GSK3640254 |
| <b>Effective Date</b> | : | 15-Jan-2020 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209713.
- This RAP is intended to describe the full analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 4 |
| 2. | SUMN<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION | 4<br>4<br>6 |
| 3. | PLAN<br>3.1. | NED ANALYSESFinal Analyses | |
| 4. | ANAL<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 9<br>9 |
| 6. | STUD<br>6.1. | Y POPULATION ANALYSES Overview of Planned Study Population Analyses | |
| 7. | PHAR 7.1. | Primary Pharmacokinetic Analyses 7.1.1. Endpoint / Variables 7.1.1.1. Drug Concentration Measures 7.1.1.2. Derived Pharmacokinetic Parameters. 7.1.2. Summary Measure 7.1.3. Population of Interest 7.1.4. Statistical Analyses / Methods 7.1.4.1. Statistical Methodology Specification Secondary Pharmacokinetic Analyses 7.2.1. Endpoint / Variables | 12<br>12<br>12<br>12<br>13<br>13 |
| 8. | QAEE. | 7.2.1.1. Drug Concentration Measures 7.2.1.2. Derived Pharmacokinetic Parameters 7.2.2. Summary Measure 7.2.3. Population of Interest 7.2.4. Statistical Analyses / Methods | 14<br>15<br>15 |
| 0. | 8.1.<br>8.2.<br>8.3.<br>8.4. | Adverse Events Analyses | 16<br>16<br>16 |

209713

| 9. | REFE | RENCES. | | 18 |
|---|---|---|---|---|
| 10. | APPE | NDICES | | 19 |
| | 10.1. | | x 1: Schedule of Activities | |
| | | | Protocol Defined Schedule of Events | |
| | 10.2. | Appendix | c 2: Study Phases and Treatment Emergent Adverse | |
| | | | Other Other family by Flactor and State and With Cines | |
| | | 10.2.1. | | |
| | | 40.00 | 10.2.1.1. Study Phases for Concomitant Medication | 22 |
| | 40.0 | 10.2.2. | Treatment Emergent Flag for Adverse Events | 23 |
| | 10.3. | Appendix | x 3: Data Display Standards & Handling Conventions | 24 |
| | | 10.3.1.<br>10.3.2. | Reporting Process | |
| | | 10.3.2. | Reporting Standards Reporting Standards for Pharmacokinetics | |
| | 10.4. | | k 4: Derived and Transformed Data | ∠3<br>27 |
| | 10.4. | 10.4.1. | General | |
| | | 10.4.1. | Study Population | |
| | | 10.4.2. | Safety | |
| | 10.5. | | s 5: Reporting Standards for Missing Data | |
| | 10.5. | 10.5.1. | | |
| | | 10.5.1. | Handling of Missing Data | |
| | | 10.0.2. | 10.5.2.1. Handling of Missing and Partial Dates | |
| | 10.6. | Appendix | k 6: Division of AIDS (DAIDS) Table for Grading the | 20 |
| | | | of Adult and Pediatric Adverse Events | 30 |
| | | | Laboratory Values | |
| | 10.7. | | x 7: Values of Potential Clinical Importance | |
| | | | ECG | |
| | | | Vital Signs | |
| | 10.8. | | c 8: Abbreviations & Trade Marks | |
| | | 10.8.1. | Abbreviations | 34 |
| | | 10.8.2. | Trademarks | 35 |
| | 10.9. | Appendix | c 9: List of Data Displays | 36 |
| | | 10.9.1. | Data Display Numbering | 36 |
| | | 10.9.2. | Mock Example Shell Referencing | 36 |
| | | 10.9.3. | Deliverables | |
| | | 10.9.4. | Study Population Tables | |
| | | 10.9.5. | Safety Tables | |
| | | 10.9.6. | Safety Figures | 40 |
| | | 10.9.7. | Pharmacokinetic Tables | |
| | | 10.9.8. | ICH Listings | |
| | | 10.9.9. | Non-ICH Listings | 45 |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 209713.

Due to a potential contamination issue in the study drug, the study was early terminated. Only an abbreviated set of outputs will be generated to support the clinical study report.

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

This is a Phase 1, randomized, open-label, single-dose, 4-period crossover study to compare the relative bioavailability (BA) of a tablet formulation of GSK3640254 with the capsule formulation and to assess the effect of food on the pharmacokinetics (PK) of the tablet formulation in healthy participants.

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| • None | Randomized population is<br>defined as all participants<br>who were randomly<br>assigned to a treatment<br>sequence | This is a randomized study<br>and listing of randomization<br>schedule will be produced<br>based on randomized<br>population. |
| Pharmacokinetic concentration population will be used for the PK concentration listings, summary tables, and plotting of concentration-time data. | Pharmacokinetic concentration population will be used for the PK concentration listings and summary tables. | Study terminated earlier due to potential contamination issue. An abbreviated clinical study report will be reported, and PK figures are not needed. |

# 2.2. Study Objective(s) and Endpoint(s)

| Ob | pjectives | Endpoints |
|---|---|---|
| Pri | imary Objectives | Primary Endpoints |
| • | To assess the relative BA of GSK3640254 mesylate tablets and GSK3640254 mesylate capsules (in the presence of a moderate fat meal) | AUC(0-∞), AUC(0-t), Cmax, and Tmax for<br>GSK3640254 |
| • | To assess the effect of food (fasted, moderate fat meal, and high fat meal) on the PK of the GSK3640254 mesylate tablet formulation | |

209713

| Objectives | Endpoints |
|---|---|
| Secondary Objectives | Secondary Endpoints |
| To assess the safety and tolerability of GSK3640254 following single oral administration to healthy participants under fasted or fed (moderate fat or high fat) conditions | Safety and tolerability parameters for<br>AEs/SAEs, observed and change from<br>baseline clinical laboratory assessments,<br>ECGs, and vital sign measurements |
| To characterize the PK of GSK3640254 | <ul><li>tlag, t1/2, CL/F, and Vz/F for GSK3640254</li><li>GSK3640254 PK concentrations in plasma</li></ul> |

AE = adverse event;  $AUC(0-\infty)$  = area under the plasma concentration-time curve from time zero extrapolated to infinity; AUC(0-t) = area under the plasma concentration-time curve from time zero to time t; BA = bioavailability; CL/F = apparent oral clearance; Cmax = maximum observed concentration; ECG = electrocardiogram; PK = pharmacokinetics; SAE = serious adverse event; t1/2 = apparent terminal phase half-life; tlag = lag time for absorption; Tmax = time of maximum observed concentration; Vz/F = apparent volume of distribution.

### 2.3. Study Design



# 2.4. Statistical Hypotheses

There is no formal research hypothesis that will be statistically tested in this study.

# 3. PLANNED ANALYSES

### 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) have been declared by Data Management.

The study early terminated due to potential contamination issue in study drug. All participants completed Treatment Period 2 before the study was terminated.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>All participants who signed the informed consent form</li> <li>This population will be used for screen failure listing and summary.</li> </ul> | Study Population |
| Randomized | <ul> <li>All participants who were randomly assigned to a treatment sequence.</li> <li>This population will be used for listing of randomization schedule.</li> </ul> | Study Population |
| Safety | <ul> <li>All participants who received at least 1 dose of study medication.</li> <li>This population will be used for all demographic, disposition (exclude screen failure), and safety listings, summaries, and figures</li> </ul> | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>Concentration | <ul> <li>All participants who underwent plasma PK sampling and had evaluable PK assay results.</li> <li>This population will be used for the PK concentration listings and summary tables.</li> </ul> | PK Concentration |
| Pharmacokinetic<br>Parameter | <ul> <li>All participants who underwent plasma PK sampling and had evaluable PK parameters estimated.</li> <li>This population will be used for PK parameter listings, summary tables, and statistical analysis tables.</li> </ul> | <ul><li>PK Parameter</li><li>PK statistical analysis</li></ul> |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarized and listed

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan. The "significant" protocol deviation in the Protocol Deviation Management Plan is equivalent to "important" protocol deviations.

209713

- Data will be reviewed prior to freezing the database to ensure all significant deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | |
|---|---|---|
| Data Displays for Repo | Data Displays for Reporting | |
| Description | Code | Order in TLF |
| GSK3640254 200 mg (single dose given as 2 × 100-mg capsules) administered under moderate fat condition | Treatment A | 1 |
| GSK3640254 200 mg (single dose given as 2 × 100-mg tablets) administered under moderate fat conditions | Treatment B | 2 |
| GSK3640254 200 mg (single dose given as 2 × 100-mg tablets) administered under fasted conditions | Treatment C | 3 |
| GSK3640254 200 mg (single dose given as 2 × 100-mg tablets) administered under high fat condition | Treatment D | 4 |

### 5.2. Baseline Definitions

For vital signs and 12-lead ECGs, the baseline value will be the average (for quantitative assessments) or the worst case (for interpretation) of the triplicate predose assessments within each period. For clinical laboratory parameters, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. If time is not collected, Day 1 assessments within each period are assumed to be taken prior to the dose and used as baseline.

| Parameter | Study Assessments Considered as<br>Baseline | | | Baseline Used in Data Display |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | , |
| Safety | | | | |
| Vital Sign | Х | Х | X | Day 1 (Pre-Dose)[1] for each period |
| 12-Lead ECG | Χ | Х | X | Day 1 (Pre-Dose)[1] for each period |
| Hematology | Χ | Х | | Day -1 |
| Clinical<br>Chemistry | Х | Х | | Day -1 |
| Urinalysis | Х | Х | | Day -1 |

ECG = Electrocardiogram.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

<sup>[1]</sup> The average (for quantitative assessments) or the worst case (for interpretation) of the predose triplicate assessments will be used as the baseline.

209713

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Schedule of Activities |
| 10.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Reporting Standards for Missing Data |
| 10.6 | Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

209713

# 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety or Screened or Randomized population, unless otherwise specified.

Study population analyses including analyses of randomization schedule, participant disposition, protocol deviations (including inclusion/exclusion criteria deviations), demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

### 7. PHARMACOKINETIC ANALYSES

### 7.1. Primary Pharmacokinetic Analyses

### 7.1.1. Endpoint / Variables

### 7.1.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetics). Plasma concentrations of GSK3640254 will be measured and presented in tabular form and will be summarized descriptively. Plasma GSK3640254 concentration-time data will be listed by participant, treatment group and sampling time and summarized by treatment group and sampling time for each period of the study.

### 7.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits. Subjects who experience emesis at or before 2 times median  $T_{max}$  will be excluded from the calculation of summary statistics and statistical analysis for the respective treatment.

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the plasma concentration-time curve from time 0 extrapolated to infinity, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-t) | Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time of maximum observed concentration |

#### NOTES:

Additional parameters may be included as required.

# 7.1.2. Summary Measure

Pharmacokinetic parameters AUC(0- $\infty$ ), AUC(0-t), Cmax, and Tmax following single dose administration of GSK3640254 to healthy participants.

### 7.1.3. Population of Interest

The primary PK analyses will be based on the PK concentration population for plasma PK concentrations and the PK parameter population for plasma PK parameters and statistical analysis.

### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarized using descriptive statistics and listed.

Primary plasma PK parameters (AUC[0-∞], AUC[0-t], Cmax, and Tmax) will be estimated for GSK3640254. Summary statistics (arithmetic mean, geometric mean, median, standard deviation (SD), coefficient of variation (CV), minimum, maximum, between-subject coefficient of variation (CVb), and 90% confidence interval (CI) for plasma GSK3640254 PK parameter values will be summarized by treatment.

#### 7.1.4.1. Statistical Methodology Specification

The following PK statistical analyses will only be performed if sufficient data are available (i.e. if participants have well defined plasma profiles).

### **Endpoint / Variables**

 Plasma primary PK endpoints include AUC(0-∞), AUC(0-t), Cmax, and Tmax for GSK3640254 as data permit

### **Model Specification**

- Analysis will be performed to compare the relative BA of a tablet formulation of GSK3640254 with the capsule formulation, as appropriate. Analyses will be performed on the natural logarithms of AUC(0-∞), AUC(0-t), and Cmax using linear mixed-effect models with treatment, period, and sequence as fixed effects and participant as a random effect. Effects will be estimated, and CIs will be constructed for the following treatment comparisons:
  - Treatment B (test) versus Treatment A (reference)
  - Point estimates and 90% CIs for treatment differences on the log scale derived from the model will be exponentiated to obtain estimates for geometric mean ratios and CIs on the original scale.
- The effect of food (moderate or high fat meal) on the PK of the tablet formulation of GSK3640254 will be similarly analyzed for the following treatment comparisons:
  - Treatment B (test) versus Treatment C (reference)
  - Treatment D (test) versus Treatment C (reference)
- Non-parametric analysis will be performed to compare the Tmax of a tablet formulation of GSK3640254 with the capsule formulation, as appropriate. The Hodges-Lehmann estimate will be used to produce the median, median difference, and 90% CIs for the following treatment comparison:
  - Treatment B (test) versus Treatment A (reference)
  - A p-value will be generated by the Wilcoxon signed-rank test
- The effect of food (moderate or high fat meal) on the Tmax of the tablet formulation of GSK3640254 will be similarly analyzed for the following treatment comparisons:
  - Treatment B (test) versus Treatment C (reference)

Treatment D (test) versus Treatment C (reference)

### **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

- Statistical analysis for comparison of relative BA by analysis of variance (ANOVA) will be presented in tabular format with geometric mean ratios for the following treatment comparison:
  - Treatment B (test) versus Treatment A (reference)
- Statistical analysis for the effect of food (moderate or high fat meal) by ANOVA will be presented in tabular format with geometric mean ratios for the following treatment comparisons:
  - Treatment B (test) versus Treatment C (reference)
  - Treatment D (test) versus Treatment C (reference)
- Statistical analysis for comparison of Tmax of a tablet formulation with a capsule formulation by non-parametric analysis will be presented in tabular format with the median, median difference, and 90% CIs along with a p-value generated by the Wilcoxon signed-rank test for the following treatment comparison:
  - Treatment B (test) versus Treatment A (reference)
- Statistical analysis for comparison of the effect of food (moderate or high fat meal) on the Tmax by non-parametric analysis will be presented in tabular format with the median, median difference, and 90% CIs along with a p-value generated by the Wilcoxon signed-rank test for the following treatment comparisons:
  - Treatment B (test) versus Treatment C (reference)
  - Treatment D (test) versus Treatment C (reference)

# 7.2. Secondary Pharmacokinetic Analyses

### 7.2.1. Endpoint / Variables

### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic).

#### 7.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher). All calculations of non-compartmental parameters will be based on actual sampling times.

Plasma pharmacokinetic parameters listed below will be determined from the plasma concentration-time data, as data permits:

| Parameter | Parameter Description |
|-----------|-----------------------------------|
| tlag | Lag time for absorption |
| t1/2 | Apparent terminal phase half-life |
| CL/F | Apparent oral clearance |
| Vz/F | Apparent volume of distribution |

#### NOTES:

• Additional parameters may be included as required.

### 7.2.2. Summary Measure

Pharmacokinetic parameters tlag, t1/2, CL/F, and Vz/F following single dose administration of GSK3640254 to healthy participants.

### 7.2.3. Population of Interest

The secondary PK analyses will be based on the PK concentration population for plasma PK concentrations, and the PK parameter population for plasma PK parameters, unless otherwise specified.

### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.1 will be summarized using descriptive statistics and listed.

Secondary plasma PK parameters (tlag, t1/2, CL/F, and Vz/F) will be estimated for GSK3640254. Summary statistics (arithmetic mean, geometric mean, median, CV, SD, minimum, maximum, CVb, and 90% CI) for secondary plasma PK parameters of GSK3640254 will be summarized by treatment.

Summary statistics (arithmetic mean, median, standard deviation, minimum, maximum, and coefficient of variation) for plasma GSK3640254 PK concentrations will be summarized by treatment using the PK Concentration Population.

### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population unless otherwise specified.

### 8.1. Adverse Events Analyses

Adverse event analyses including the analysis of AEs, SAEs, and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards and will be graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 2.1, July 2017). The details of the planned displays are in Appendix 9: List of Data Displays.

# 8.3. Adverse Events of Special Interest

At the end of the study, QT prolongation, gastrointestinal intolerability/toxicity, psychiatric events, and nervous system disorders will be summarized by treatment. A listing will also be provided accordingly.

QT prolongation AE of special interest will be defined as cardiac disorders system organ class (SOC) plus preferred terms (PTs) using the Medical Dictionary for Regulatory Activities (MedDRA) Standardized MedDRA Query (SMQ) "Torsade de pointes/QT Prolongation" (narrow and broad terms) plus seizure.

Gastrointestinal intolerability/toxicity AEs of special interest will be defined within three narrow sub-SMQs [Gastrointestinal nonspecific symptoms and therapeutic procedures SMQ; Gastrointestinal nonspecific dysfunction SMQ; Gastrointestinal nonspecific inflammation (SMQ)] plus a selection of relevant broad PTs from the Gastrointestinal non-specific symptoms and therapeutic procedures SMQ.

Psychiatric AEs of special interest will be defined within the following:

- Sub-SMQ "Suicide/self-injury" (SMQ) from parent SMQ of "Depression and Suicide/Self Injury". Only narrow terms from the sub-SMQ selected.
- Sub-SMQ "Depression (excluding suicide and self-injury)" (SMQ) from parent SMQ of "Depression and Suicide/Self Injury". Only narrow terms from the sub-SMQ selected.
- All preferred terms from high level group term (HLGT) "Manic and Bipolar mood disorders and disturbances" under SOC "Psychiatric disorders".
- Narrow terms from SMQ "Psychosis and psychotic disorders" selected.
- All preferred terms from HLGT "Anxiety disorders and symptoms", under SOC 'Psychiatric disorders'.

209713

• All preferred terms from HLGT "Sleep Disorders and Disturbances" and HLGT "Sleep disturbances (incl subtypes)".

Nervous system disorders AEs of special interest will be defined within the following:

• Four HLGTs under Nervous System Disorders SOC: "Headaches"; "Mental impairment disorders"; "Neurological disorders" and "Seizures"

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including electrocardiograms (ECGs), and vital signs will be based on GSK Core Data Standards, unless otherwise specified. A figure of mean change from baseline in QTc using the Fridericia formula (QTcF) interval along with the 2-sided 95% CI using Student's t distribution will be presented by treatment and visit. The details of the planned displays are presented in Appendix 9: List of Data Displays.

209713

# 9. REFERENCES

ViiV Healthcare group of companies Document Number 2018N383392\_00 (30-AUG-2019): A Randomized, Open-Label, Single Dose, Four-Period Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants.

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Schedule of Events

# **Screening Visit**

| Procedure | Screening (up to 28 days before Day 1) |
|---|---|
| Outpatient visit | Χ |
| Informed consent | X |
| Inclusion and exclusion criteria | X |
| Demography | X |
| Full physical examination including height and weight <sup>1</sup> | X |
| Laboratory assessments (hematology, chemistry, urinalysis) | X |
| 12-lead electrocardiogram | X |
| Vital sign measurements | X |
| Medication/drug/alcohol history | X |
| Past and current medical conditions | X |
| Columbia Suicide Severity Rating Scale | X |
| Serum pregnancy test | X |
| Follicle-stimulating hormone (as needed, to confirm postmenopausal status) | Х |
| Drug, alcohol, and cotinine screen | X |
| Human immunodeficiency virus, hepatitis B and C Screening | Х |

<sup>1.</sup> A full physical examination will include at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal (GI), and neurological systems.

209713

# **Time and Events Table**

| Procedure | Check-in | | Periods | 1, 2, and 3 | } | | Perio | d 4 only | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Davis | Davi | | Washou | ıt | Davis | Davis | D | D |
| | | Day<br>1 | Day<br>2 | Days<br>3-5 | Days<br>6-7 | Day<br>1 | Day<br>2 | Days<br>3-4 | Day<br>5⁰ | |
| Admit to clinic | Х | | | | | | | | | |
| Discharge from clinic | | | | | | | | | Х | Discharge from clinic following completion of the last study procedure on Day 5 of Period 4. |
| Brief physical examination | X | | | | D7<br>(Period 2<br>only) | | | | Х | Interim or symptom targeted physical examination will be performed at the discretion of the investigator. See Protocol Section 8.2.1 for description of brief physical examination. |
| Vital signs | Х | Х | Х | D3-5 | | Х | Х | Х | Х | Blood pressure and pulse will be measured in triplicate predose on Day 1 in Periods 1-4. Single blood pressure and pulse will be measured predose on other study days. |
| 12-lead ECG | X | Х | | | | Х | | | Х | All ECGs on Day 1 in Periods 1-4 will be predose, postdose at 2 hours, and postdose at 4 hours. The predose ECGs in Periods 1-4 will be taken in triplicate. |
| Drug, alcohol, and cotinine screen | Х | | | | | | | | | See Protocol Appendix 2 for specific tests to be performed. |
| Laboratory<br>assessments<br>(hematology, chemistry,<br>urinalysis) | Х | | Х | | | | Х | | Х | See Protocol Appendix 2 for specific tests to be performed. Day 2 samples in each period to be collected 24 hours after dosing. |
| Pregnancy test | Х | | | | | | | | Х | Serum testing at Day -1 |

209713

| Procedure | Check-in | Check-in Periods 1, 2, and 3 | | | | | Perio | d 4 only | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day<br>–1 | | D | | Washou | t | D | Davi | D | Davis |
| | | Day<br>1 | Day<br>2 | Days<br>3-5 | Days<br>6-7 | Day<br>1 | Day<br>2 | Days<br>3-4 | Day<br>5º | |
| Columbia-Suicide<br>Severity<br>Rating Scale | Х | | | | D7 | | | | Х | |
| Genetic sample (optional) | Х | | | | | | | | | |
| Study intervention:<br>GSK3640254 200 mg<br>(capsule or tablet) | | Х | | | | х | | | | Participants will fast overnight for at least 10 hours prior to dosing; be provided a moderate fat meal, a high fat meal, or no meal 30 minutes prior to dosing; and be provided standardized meals ≥4 hours postdose. See Protocol Section 4.1. |
| Serial PK sampling | | Х | Х | Х | | Х | Х | Х | Х | Blood collection for PK analysis of GSK3640254 will be collected within 40 minutes prior to dosing and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose in each period. |
| AE review | | <b>←</b> == | | | | :X====== | | | <b>&gt;</b> | |
| SAE review | <b>←</b> ==== | | | | ====X==== | | | | <b>&gt;</b> | |
| Concomitant medications | <b>←</b> ==== | ====== | ====== | | -===X==== | ======= | ======= | ======= | :=== <b>→</b> | |

AE = adverse event; D = day; ECG = electrocardiogram; PK = pharmacokinetic; SAE = serious adverse event.

1 Evaluations scheduled for Day 5 in Period 4 will also be performed for participants who discontinue early.

# 10.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

# 10.2.1. Study States for Lab, Electrocardiograms, and Vital Signs

Assessments and events will be classified according to the time of occurrence relative to study treatment start date(/time) and stop date(/time).

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date and Time ≤ Study Treatment Start Date and Time |
| On-Treatment | Study Treatment Start Date and Time < Date and Time ≤ Study Treatment Stop Date and Time + 5 days the Date and Time of Early Withdrawal Visit whichever is later. |
| Post-Treatment | Date and Time > Study Treatment Stop Date and Time + 5 days or the Date and Time of Early Withdrawal Visit whichever is later |

### 10.2.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|-------------|------------------------------------------------------------|
| Prior | If medication end date is not missing and is before Day -1 |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

209713

# 10.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date and time is on or after treatment start date and time &amp; on or before treatment stop date and time + 5 days.</li> <li>Study Treatment Start Date and Time ≤ AE Start Date and Time ≤ Study Treatment Stop Date and Time + 5 days.</li> <li>If the AE onset date is completely missing, the AE is considered as treatment emergent.</li> </ul> |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for adverse events. Use the rules in this table if the adverse event onset date is completely missing.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

### 10.3.1. Reporting Process

| Software | |
|---|---|
| The currently sup | The currently supported versions of SAS software (9.4) will be used. |
| Reporting Area | |
| HARP Server | \\us1salx00259.corpnet2.com |
| HARP Compound | GSK3640254 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1).</li> </ul> | |
| <ul> <li>For creation of ADaM datasets (ADC1/ADCM/ADAE), the same version of dictionary datasets will be</li> </ul> | |

### **Generation of RTF Files**

• RTF files will be generated for all reporting efforts described in the RAP.

implemented as those being used for conversion from SI to SDTM.

### 10.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK CSR. All participant level listings should be located in the modular appendices as ICH or non-ICH listings.

#### **Formats**

- All data will be reported according to the actual treatment the participant received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures, and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).

- Unscheduled or unplanned readings will be presented within the participant's listings.
- Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be
  included in listings but omitted from figures (mean figures only for PK concentrations), summaries,
  and statistical analyses (excluding statistical analyses of PK parameters).

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables except for determining the worst-case values.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | <u> </u> |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 10.3.3. Reporting Standards for Pharmacokinetics

| TOIOIOI TROPOI | ang standards for Friatmassianistics |
|---|---|
| Pharmacokinetic Con | centration Data |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | <ul> <li>Refer to IDSL PK Display Standards.</li> <li>Refer to IDSL Statistical Principle 6.06.1.</li> <li>For continuous data: <ul> <li>NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.</li> <li>For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);</li> <li>for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)</li> <li>for summary statistics, these are set to 0 (to avoid skewing of the</li> </ul> </li> </ul> |
| | <ul> <li>summary statistics)</li> <li>Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly)</li> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> <li>Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only.</li> </ul> |
| Pharmacokinetic Parameter Data | |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | N, n, arithmetic mean, 90% CI of arithmetic mean, geometric mean, 95% CI of geometric mean, SD, SD of logged data CV (%), and between-subject geometric coefficient of variation (CVb (%)) will be reported. CV <sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of Ln-Transformed data) |

# 209713 | Statistical Analysis Plan RAP 15 Jan 2020 | TMF-1623402 | 2.0

# CONFIDENTIAL

209713

| Parameters Not<br>Being Ln-<br>Transformed | Tmax, tlag, λz, λz lower, λz upper, and λz no. of points. |
|---|---|
| Parameters Not<br>Being Summarized | λz, λz lower, λz upper, and λz no. of points. |
| Listings | Include the first point, last point and number of points used in the determination of $\lambda z$ and Rsq_adjusted for listings. |

209713

### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- The worst finding/interpretation associated with multiple measurements as the finding/interpretation for that time point.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from Dose Date on Period 1 Day 1:
  - Assessment Date = Missing
    - → Study Day = Missing
  - Assessment Date < Dose Date on Period 1 Day 1</li>
    - → Study Day = Assessment Date –Dose Date on Period 1 Day 1
  - Assessment Date >= Dose Date on Period 1 Day 1
    - → Study Day = Assessment Date Dose Date on Period 1 Day 1 + 1

#### **Period Day**

- Calculated as the number of days from First Dose Date for the respective period:
  - Assessment Date = Missing
    - → Period Day = Missing
  - Assessment Date < Dose Date on Period 1 Day 1</li>
    - → Period Day = Assessment Date Dose Date on Period 1 Day 1
  - Dose Date on Period 1 Day 1 <= Assessment Date < Dose Date on Period 2 Day 1</li>
    - → Period Day = Assessment Date Dose Date on Period 1 Day 1 + 1
  - Dose Date on Period 2 Day 1 <= Assessment Date < Dose Date on Period 3 Day 1</li>
    - → Period Day = Assessment Date Dose Date on Period 2 Day 1 + 1
  - Dose Date on Period 3 Day 1 <= Assessment Date < Dose Date on Period 4 Day 1</li>
    - → Period Day = Assessment Date Dose Date on Period 3 Day 1 + 1
  - Assessment Date >= Dose Date on Period 4 Day 1
    - → Period Day = Assessment Date Dose Date on Period 4 Day 1 + 1

# 10.4.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - o Any participant with a missing day and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

209713

### 10.4.3. Safety

# Adverse Events

# **AEs of Special Interest**

- QT prolongation
- Gastrointestinal intolerability/toxicity
- Psychiatric events
- Nervous system disorders

### 12-Lead Electrocardiograms

### **QTcB** Interval

 QTc using the Bazett formula (QTcB) interval in msec will be calculated using QT interval (msec) and RR (msec) as

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

where RR interval in msec is calculated using QT interval (msec) and QTcF interval (msec) as

$$RR = (\frac{QT}{QTcF})^3 \times 1000$$

# 10.5. Appendix 5: Reporting Standards for Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as the participant had completed all phases of the study including the final date on which data were or are expected to be collected.</li> <li>Withdrawn participants were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the CSR. |

# 10.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

209713

# 10.6. Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

# 10.6.1. Laboratory Values

Laboratory abnormalities will be graded according to the DAIDS grading table Version 2.1, July 2017. Laboratory results are converted to use SI units; only the numeric part of the criteria will be used. If for a laboratory parameter there are multiple grades sharing the same criteria, the maximum grade will be used.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Lymphocyte Count, Low (cell/mm³; cells/L) > 5 years of age (not HIV infected) | 600 to < 650<br>0.600 × 10 <sup>9</sup> to < 0.650 × 10 <sup>9</sup> | 500 to < 600<br>0.500 × 10 <sup>9</sup> to < 0.600 ×<br>10 <sup>9</sup> | 350 to < 500<br>0.350 × 10 <sup>9</sup> to < 0.500 × 10 <sup>9</sup> | < 350<br>< 0.350 × 10 <sup>9</sup> |
| Absolute Neutrophil Count, Low (cells/mm³; cells/L) > 7 days of age | 800 to 1,000<br>0.800 × 10 <sup>9</sup> to 1.000 × 10 <sup>9</sup> | 600 to 799<br>0.600 × 10 <sup>9</sup> to 0.799 ×<br>10 <sup>9</sup> | 400 to 599<br>0.400 × 10 <sup>9</sup> to 0.599 × 10 <sup>9</sup> | < 400<br>< 0.400 × 10 <sup>9</sup> |
| Hemoglobin, Low (g/dL; mmol/L) | 10.0 to 10.9 | 9.0 to < 10.0 | 7.0 to < 9.0 | < 7.0 |
| ≥ 13 years of age (male only) | 6.19 to 6.76 | 5.57 to < 6.19 | 4.34 to < 5.57 | <4.34 |
| Hemoglobin, Low (g/dL; mmol/L) | 9.5 to 10.4 | 8.5 to < 9.5 | 6.5 to < 8.5 | < 6.5 |
| ≥ 13 years of age (female only) | 5.88 to 6.48 | 5.25 to < 5.88 | 4.03 to < 5.25 | < 4.03 |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to < 125,000<br>100.000 × 10 <sup>9</sup> to < 125.000<br>× 10 <sup>9</sup> | 50,000 to < 100,000<br>50.000 × 10 <sup>9</sup> to <<br>100.000 × 10 <sup>9</sup> | 25,000 to < 50,000<br>25.000 × 10 <sup>9</sup> to < 50.000 ×<br>10 <sup>9</sup> | < 25,000<br>< 25.000 × 10 <sup>9</sup> |
| White Blood Cell, Decreased (cells/mm³; cells/L) > 7 days of age | 2,000 to 2,499<br>2.000 × 10 <sup>9</sup> to 2.499 × 10 <sup>9</sup> | 1,500 to 1,999<br>1.500 × 10 <sup>9</sup> to 1.999 ×<br>10 <sup>9</sup> | 1,000 to 1,499<br>1.000 × 109 to 1.499 × 109 | < 1,000<br>< 1.000 × 10 <sup>9</sup> |

209713

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Albumin, Low (g/dL; g/L) | 3.0 to < LLN<br>30 to < LLN | ≥ 2.0 to < 3.0<br>≥ 20 to < 30 | < 2.0<br>< 20 | NA |
| Alkaline Phosphatase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 × ULN |
| Alanine Aminotransferase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 ULN |
| Amylase (Total), High | 1.1 to < 1.5 × ULN | 1.5 to < 3.0 × ULN | 3.0 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Aspartate Aminotransferase, High | 1.25 to < 2.5 × ULN | 2.5 to < 5.0 × ULN | 5.0 to < 10.0 × ULN | ≥ 10.0 × ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to < LLN<br>16.0 to < LLN | 11.0 to < 16.0<br>11.0 to < 16.0 | 8.0 to < 11.0<br>8.0 to < 110. | < 8.0<br>< 8.0 |
| Direct Bilirubin, High > 28 days of age | NA | NA | > ULN with other signs and symptoms of hepatotoxicity | > ULN with life-threatening consequences (e.g., signs and symptoms of liver failure) |
| Total Bilirubin, High > 28 days of age | 1.1 to < 1.6 × ULN | 1.6 to < 2.6 × ULN | 2.6 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Calcium, High (mg/dL; mmol/L) | 10.6 to < 11.5 | 11.5 to < 12.5 | 12.5 to < 13.5 | ≥ 13.5 |
| ≥ 7 days of age | 2.65 to < 2.88 | 2.88 to < 3.13 | 3.13 to < 3.38 | ≥ 3.38 |
| Calcium, Low (mg/dL; mmol/L) | 7.8 to < 8.4 | 7.0 to < 7.8 | 6.1 to < 7.0 | < 6.1 |
| ≥ 7 days of age | 1.95 to < 2.10 | 1.75 to < 1.95 | 1.53 to < 1.75 | < 1.53 |
| Creatine Kinase, High | 3 to < 6 × ULN | 6 to < 10 × ULN | 10 to < 20 × ULN | ≥ 20 × ULN |
| Creatinine, High Choose the method that selects for the higher grade | 1.1 to 1.3 × ULN | > 1.3 to 1.8 × ULN OR<br>Increase to 1.3 to < 1.5 ×<br>participant's baseline | > 1.8 to < 3.5 ULN OR<br>Increase to 1.5 to < 2.0 ×<br>participant's baseline | ≥ 3.5 × ULN OR Increase of ≥ 2.0 × participant's baseline |
| Glucose Fasting, High (mg/dL; mmol/L) | 110 to 125<br>6.11 to < 6.95 | > 125 to 250<br>6.95 to < 13.89 | > 250 to 500<br>13.89 to < 27.75 | ≥ 500<br>≥ 27.75 |
| Glucose, Low (mg/dL; mmol/L) | 55 to 64 | 40 to < 55 | 30 to < 40 | < 30 |
| ≥ 1 month of age | 3.05 to < 3.55 | 2.22 to < 3.05 | 1.67 to < 2.22 | < 1.67 |
| Lipase, High | 1.1 to < 1.5 × ULN | 1.5 to < 3.0 × ULN | 3.0 to < 5.0 × ULN | ≥ 5.0 × ULN |
| Cholesterol, Fasting, High (mg/dL;<br>mmol/L)<br>≥ 18 years of age | 200 to < 240<br>5.18 to < 6.19 | 240 to < 300<br>6.19 to < 7.77 | ≥ 300<br>≥ 7.77 | NA |
| Triglycerides, Fasting, High (mg/dL; | 150 to 300 | > 300 to 500 | > 500 to < 1.000 | > 1,000 |
| mmol/L) | 1.71 to 3.42 | > 3.42 to 5.7 | > 5.7 to 11.4 | > 11.4 |
| Phosphate, Low (mg/dL; mmol/L) > 14 years of age | 2.0 to < LLN<br>0.65 to < LLN | 1.4 to < 2.0<br>0.45 to < 0.65 | 1.0 to < 1.4<br>0.32 to < 0.45 | < 1.0<br>< 0.32 |

209713

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Potassium, High (mEq/L; mmol/L) | 5.6 to < 6.0 | 6.0 to < 6.5 | 6.5 to < 7.0 | ≥ 7.0 |
| | 5.6 to < 6.0 | 6.0 to < 6.5 | 6.5 to < 7.0 | ≥ 7.0 |
| Potassium, Low (mEq/L; mmol/L) | 3.0 to < 3.4 | 2.5 to < 3.0 | 2.0 to < 2.5 | < 2.0 |
| | 3.0 to < 3.4 | 2.5 to < 3.0 | 2.0 to < 2.5 | < 2.0 |
| Sodium, High (mEq/L; mmol/L) | 146 to < 150 | 150 to < 154 | 154 to < 160 | ≥ 160 |
| | 146 to < 150 | 150 to < 154 | 154 to < 160 | ≥ 160 |
| Sodium, Low (mEq/L; mmol/L) | 130 to < 135 | 125 to < 130 | 121 to < 125 | ≤ 120 |
| | 130 to < 135 | 125 to < 130 | 121 to < 125 | ≤ 120 |
| Uric Acid, High (mEq/L; mmol/L) | 7.5 to < 10.0 | 10.0 to < 12.0 | 12.0 to < 15.0 | ≥ 15.0 |
| | 0.45 to < 0.59 | 0.59 to < 0.71 | 0.71 to < 0.89 | ≥ 0.89 |

NA=not applicable; LLN = lower limit of normal; ULN=upper limit of normal.

| Urinalysis | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Glucose/Glycosuria (random collection tested by dipstick) | Trace to 1+ or ≤ 250 mg | 2+ or > 250 to ≤ 500 mg | > 2+ or > 500 mg | NA |
| Protein/Proteinuria (random collection tested by dipstick) | 1+ | 2+ | 3+ or higher | NA |
| Red Blood Cells (RBCs)/Hematuria (not<br>to be reported based on dipstick findings<br>or on blood believed to be of menstrual<br>origin) | 6 to < 10 RBCs per high<br>power field | ≥ 10 RBCs per high power field | Gross, with or without clots<br>OR with RBC casts OR<br>intervention indicated | Life-threatening consequences |

NA=not applicable

209713

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. ECG

| ECG Parameter | Units | Potential Clinically | Potential Clinically Important Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | • | | |
| Absolute QTc Interval | msec | <320 | >450 |
| Absolute PR Interval | msec | < 120 | > 200 |
| Absolute QRS Interval | msec | < 60 | > 120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 10.7.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically | Important Range |
|--------------------------|-------|----------------------|-----------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 140 |
| Diastolic Blood Pressure | mmHg | < 45 | > 90 |
| Heart Rate | bpm | < 40 | > 100 |

209713

# 10.8. Appendix 8: Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|-----------------|------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ANOVA | Analysis of Variance |
| AUC | Area under the Plasma Concentration-Time Curve |
| AUC(0-∞) | AUC from Time 0 Extrapolated to Infinity |
| AUC(0-t) | AUC from Time 0 to Time t |
| BA | Bioavailability |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | Apparent Oral Clearance |
| Cmax | Maximum Observed Concentration |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CV | Coefficient of Variation |
| CV <sub>b</sub> | Coefficient of Variation (Between) |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| HLGT | High Level Group Term |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| LLN | Lower Limit of Normal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QTcB | QTc using the Bazett formula |
| QTcF | QTc using the Fridericia formula |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| t1/2 | Apparent Terminal Phase Half-life |
| tlag | Lag Time for Absorption |
| Tmax | Time of Maximum Observed Concentration |
| ULN | Upper Limit of Normal |

209713

| Abbreviation | Description |
|--------------|---------------------------------|
| Vz/F | Apparent Volume of Distribution |

# 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

### 10.9. Appendix 9: List of Data Displays

# 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|---------|
| Study Population | 1.1 to 1.4 | |
| Safety | 2.1 to 2.15 | 2.1 |
| Pharmacokinetic | 3.1 to 3.7 | |
| Section | Listings | |
| ICH Listings | 1 to 32 | |
| Other Listings | 33 to 34 | |

### 10.9.2. Mock Example Shell Referencing

Non-IDSL specifications will be referenced as indicated and if required example mock-up displays provided in the Table/Listing/Figure Shells.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 10.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

209713

# 10.9.4. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2. | Screened | SD1 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| Demographic and Baseline Characteristics | | | | | |
| 1.3. | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.4. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |

209713

# 10.9.5. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1CP | Summary of Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.2. | Safety | AE1CP | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.3. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.4. | Safety | AE1CP | Summary of Adverse Events of Special Interest by System Organ Class and Preferred Term | | SAC |
| Labora | tory: Chemistry | у | | | |
| 2.5. | Safety | LB1 | Summary of Clinical Chemistry Data | | SAC |
| 2.6. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | | SAC |
| Labora | tory: Hematolo | gy | | | |
| 2.7. | Safety | LB1 | Summary of Hematology Data | | SAC |
| 2.8. | Safety | LB1 | Summary of Hematology Changes from Baseline | | SAC |
| Labora | tory: Urinalysis | 3 | | | |
| 2.9. | Safety | LB1 | Summary of Urine Concentration | | SAC |
| 2.10. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | | SAC |
| ECG | | | | | |
| 2.11. | Safety | EG2 | Summary of ECG Values | | SAC |

209713

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | Safety | EG2 | Summary of ECG Changes from Baseline | | SAC |
| Vital Signs | | | | | |
| 2.13. | Safety | VS1 | Summary of Vital Signs | | SAC |
| 2.14. | Safety | VS1 | Summary of Vital Sign Changes from Baseline | | SAC |
| C-SSRS | | | | | |
| 2.15. | Safety | CSSRS4 | Listing of C-SSRS Suicidal Ideation and Behavior Data | Only include participants who have suicidal ideation or behavior | SAC |

209713

# 10.9.6. Safety Figures

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | ECG | | | | |
| 2.1. | Safety | EG9 | Mean (95% CI) Change from Baseline in QTcF Interval by Timepoint and Treatment | | SAC |

209713

# 10.9.7. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Co | ncentration Data | | | | |
| 3.1. | PK<br>Concentration | PKCT1 | Summary of GSK3640254 Plasma Pharmacokinetic Concentration-Time Data (ng/mL) by Treatment | | SAC |
| PK Dei | rived Parameters | 3 | | | |
| 3.2. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment | Parameters with units; present PK parameters in ug/mL or ug.h/mL | SAC |
| 3.3. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma<br>Pharmacokinetic Parameters (Ln-Transformed) Based on Actual<br>Time by Treatment | Parameters with units; present PK parameters in ug/mL or ug.h/mL | SAC |
| PK An | alysis Tables | | | | |
| 3.4. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA)- Relative Bioavailability | AUC(0-∞), AUC(0-t) and Cmax, | SAC |
| 3.5. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA)- Food Effect | AUC(0-∞), AUC(0-t) and Cmax, | SAC |
| 3.6. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Non-parametric analysis- Relative Bioavailability | Tmax | SAC |
| 3.7. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Non-parametric analysis-Food Effect | Tmax | SAC |

209713

# 10.9.8. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | · |
| 1. | Randomized | POP_L1 | Listing of Randomization Schedule | | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| Protoco | ol Deviations | | | | |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 5. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analyzed | | | | · |
| 6. | Safety | SP3A | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | · |
| 7. | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 8. | Safety | DM9 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | · |
| 9. | Safety | CM5 | Listing of Concomitant Medications | Based on GSK Drug Dictionary | SAC |
| Exposu | ire and Treatme | ent Compliance | | | |
| 10. | Safety | EX4 | Listing of Exposure Data | | SAC |
| 11. | Safety | POP_L2 | Listing of Meal Data | | SAC |
| Advers | Adverse Events | | | | |
| 12. | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC |

209713

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 13. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 14. | Safety | AE9CP | Listing of All Adverse Events | | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 15. | Safety | AE9CP | Listing of Study Drug Related Adverse Events | | SAC |
| 16. | Safety | AE9CP | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | SAC |
| 17. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 18. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| 19. | Safety | AE9CP | Listing of Adverse Events of Special Interest | | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| All Lab | oratory | | | 1 | |
| 22. | Safety | LB5A | Listing of Clinical Chemistry with any Toxicities | | SAC |
| 23. | Safety | LB5A | Listing of All Clinical Chemistry Data for Subjects with any Toxicities | | SAC |
| 24. | Safety | LB5A | Listing of Hematology with any Toxicities | | SAC |
| 25. | Safety | LB5A | Listing of All Hematology Data for Subjects with any Toxicities | | SAC |
| 26. | Safety | LB5A | Listing of Urinalysis with any Toxicities | | SAC |
| 27. | Safety | LB5A | Listing of All Urinalysis Data for Subjects with any Toxicities | | SAC |
| ECG | • | | | • | - ' |
| 28. | Safety | EG6 | Listing of All ECG Findings | | SAC |

209713

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 29. | Safety | EG6 | Listing of All Abnormal ECG Findings | | SAC |
| 30. | Safety | EG4 | Listing of All ECG Values | | SAC |
| Vital Si | gns | | | | |
| 31. | Safety | VS5 | Listing of All Vital Signs of Potential Clinical Importance | | SAC |
| 32. | Safety | VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

209713

# 10.9.9. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | Pharmacokinetics | | | | |
| 33. | PK<br>Concentration | PKCL1P | Listing of GSK3640254 Plasma Concentration-Time Data by Treatment | | SAC |
| 34. | PK<br>Parameter | PKPL1P | Listing of GSK3640254 Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment | | SAC |